CLINICAL TRIAL: NCT06271252
Title: A Phase I/II, Open-label, Multicenter Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of Anti-GPRC5D CAR-T Cell Product (OriCAR-017) in Subjects With Relapsed/Refractory Multiple Myeloma.
Brief Title: A Study to Evaluate the Safety, PK/PD of (OriCAR-017) in Subjects With RR/MM - RIGEL Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OriCell Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OriCAR-017-US-P1
Record Dates: First submitted 2024-01-26; First posted 2024-02-21 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases; Multiple Myeloma
Keywords: R/R MM, CAR-T
MeSH Terms: conditions — Neoplasms, Plasma Cell; Neoplasms by Histologic Type; Neoplasms; Hemostatic Disorders; Vascular Diseases; Cardiovascular Diseases; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Hemorrhagic Disorders; Lymphoproliferative Disorders; Immunoproliferative Disorders; Immune System Diseases; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OriCAR-017 (Experimental): Single OriCAR-017 infusion
  Interventions: Drug: OriCAR-017

INTERVENTIONS:
Drug: OriCAR-017 — Anti-GPRC5D CAR-T cell product

SUMMARY:
The is a first clinical study for Oricell Therapeutics Inc. in the United States to evaluate the safety, PK, PD and preliminary efficacy of our anti-GPRC5D cell product (OriCAR-017) in subjects with relapsed/refractory multiple myeloma.

RIGEL Study

DETAILED DESCRIPTION:
This is a Phase I/II, open-label multicenter study to evaluate the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of anti-GPRC5D CAR-T cell product (OriCAR-017) in subjects with relapsed/refractory multiple myeloma". The study will consist of a Phase I dose escalation stage involving three doses as a single IV infusion) with up to 18 evaluable subjects and a dose expansion stage with 10-15 evaluable subjects, followed by a Phase II stage with up to 48 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

Capable of giving signed informed consent

Subjects aged 18 to 75 years (inclusive) at Screening (signing the ICF).

Expected survival period is >12 weeks.

Diagnosis of MM according to the IMWG criteria (2016 version).

One of the following criteria must be met:

If immunoglobulin (Ig)G type MM, then serum M protein >10 g/L; if IgA, IgD, IgE or IgM type MM, then serum M protein >5 g/L

Urine M protein level >200 mg/24 hour

If light chain type MM, then serum free light chain (sFLC) >100 mg/L and K/λ FLC ratio is abnormal.

Extramedullary lesions (>1 cm for diameter of the short axis).

For Phase I (dose-escalation) - Subjects who had received at least 3 prior lines of therapy, had previous exposure to BCMA-Ag+ therapies, and were refractory to the last line of therapy.

For Phase I (dose-expansion) and Phase II: Subjects with previous exposure to BCMA directed therapies including BCMA bispecific antibody (e.g., teclistamab), BCMA antibody directed conjugate (such as BLENREP), and BCMA-CAR-T (such as CARVYKT1TM)

Subjects with adequate hematologic, renal, hepatic, pulmonary and cardiac function.

Subject and partners willing to take and or use effective contraceptive measures until 2 years post IMP infusion.

Exclusion Criteria:

Pregnant or breastfeeding.

Seropositive for history of human immunodeficiency virus Active Hepatitis B infection and or Hepatitis C infection

Known active or prior history of CNS involvement

History of autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) caused damage to terminal organs or required systemic application of immunosuppressive or other drugs in the past 2 years

Presence of uncontrolled active infection

Subjects who received autologous hematopoietic stem cell transplantation (ASCT) within 8 weeks of Screening Visit or who plan to undergo ASCT during the study.

Subjects who received allogeneic stem cell therapy.

Any condition that in the opinion of the Investigator, would interfere with evaluation of the IMP.

Received Bendamustine treatment 1 year prior to Screening Visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2026-12-12 (Estimated); Study Completion 2028-04-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of OriCAR-017 US-P1 | Up to 28 days
  The MTD is defined as the highest dose with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level.
Dose-limiting toxicity (DLT) | Up to 28 days
  A DLT is defined as any of the treatment-emergent adverse events (TEAEs; a TEAE is defined as an adverse event [AE] that starts on or after the first administration of study medication) condition or concomitant medications.

SECONDARY OUTCOMES:
Evaluate PK parameters of OriCAR-017 in subjects with relapsed/refractory MM | Up to 2 years
  Assess concentration of CAR-T cells in peripheral blood
Evaluate PD parameters of OriCAR-017 in subjects with relapsed/refractory MM | Up to 2 years
  Assess PD markers related to CAR-T therapy in peripheral blood.
Assessment of Duration of Response (DOR) of treatment in patients with RR/MM | Up to 2 years
  DOR as assessed by Local Investigators according to the IMWG Criteria
Progress-Free Survival (PFS) of treatment in patients with RR/MM | Up to 2 years
  PFS as assessed by Local Investigators according to the IMWG Criteria
Assessment of Overall Survival (OS) of treatment in patients with RR/MM | Up to 2 years
  OS as assessed by Local Investigators according to the IMWG Criteria
Assessment of MRD negative Rate | Up to 2 years
  Proportion of subjects with MRD negative status by flow cytometry
Assessment of Overall Response Rate (ORR) | Up to 2 years
  Percentage of subjects with PR, + VGPR+ CR + strict complete response (sCR) as assessed by Local Investigator according to the IMWG criteria
Assessment of Disease Control Rate (DCR) | Up to 2 years
  Percentage of subjects with CBR (Clinical Benefit Rate) + Stable Disease as assessed by Local Investigator according to IMWG Criteria
Assessment of Clinical Benefit Rate (CBR) | Up to 2 years
  Percentage of subjects with ORR + Minimal Response by Local Investigator according to IMWG Criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Northside Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No